CLINICAL TRIAL: NCT03156283
Title: SleepWell24: An Innovative Smartphone Application to Improve PAP Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Megan Petrov, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5R21NR016046-02 (NIH); R21NR016046 (NIH)
Record Dates: First submitted 2017-04-27; First posted 2017-05-17 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Obstructive Sleep Apnea of Adult
Keywords: smartphone; obstructive sleep apnea; adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Fitness Trackers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SleepWell24 Application (Experimental): A mobile health smartphone application based on evidence-based health behavior change theory and interventions to promote adherence to positive airway pressure therapy
  Interventions: Behavioral: SleepWell24 Application
- Usual Care Plus Activity Monitor (Other): Per usual clinical care standards within the Center for Sleep Medicine at Mayo Clinic Arizona, all patients will receive instructions/education on positive airway pressure (PAP) use, multiple mask fittings, encouragement to use PAP every night, and staff is available in the event of problems. Control patients will also receive a wearable activity monitor to use during the study. The wearable sensor will be used to isolate the effect of SleepWell24 on PAP adherence from potential novelty effects due to receiving a generic health behavior change app.
  Interventions: Other: Usual Care Plus Activity Monitor

INTERVENTIONS:
Behavioral: SleepWell24 Application — An evidence-based behavioral change smartphone application designed to promote adherence to positive airway pressure (PAP) therapy
  Arms: SleepWell24 Application
Other: Usual Care Plus Activity Monitor — Participants will receive usual care at the Mayo Clinic Center for Sleep Medicine when first diagnosed with sleep apnea and prescribed positive airway pressure therapy. In addition, they will receive a commercial activity monitor with an associated smartphone application to isolate the effect of SleepWell24 on PAP adherence from potential novelty effects due to receiving a generic health behavior change app.
  Arms: Usual Care Plus Activity Monitor

SUMMARY:
Obstructive sleep apnea (OSA) is a major public health concern n the United States. Positive airway pressure (PAP) therapy is the treatment-of-choice and "gold standard" for individuals with moderate-to-severe OSA. Regular and sustained PAP use can reduce risk for subsequent disease and improve quality of life. Nevertheless, PAP adherence rates are low. Most PAP adherence programs do not address the self-management skills and strategies that promote adherence and are often too costly and complex to integrate into overburdened clinical environments. Furthermore, they do not leverage opportunities to change lifestyle behaviors that occur across the 24h spectrum (i.e., sleep hygiene, sedentary behavior, physical activity), which have promise to improve OSA symptoms and PAP adherence. The investigators have previously developed and successfully tested BeWell24, a multicomponent smartphone "app" that uses evidence-based behavior change strategies to improve sleep, sedentary, and physical activity behaviors. The investigators will enhance this app to create SleepWell24. Enhancements will include: (1) specific behavior change strategies from the evidence-based Sleep Apnea Self-Management Program to promote PAP adherence; (2) an interface for exchange of patient data to facilitate patient-provider communication on treatment progress; and (3) real-time feedback via wireless integration with a consumer-based PAP machine and wearable sensor. All aspects of this work will be embedded within the Mayo Clinic Arizona Center for Sleep Medicine. The investigators will test the effects of SleepWell24 in newly prescribed PAP users and gather data on the feasibility and acceptability of using SleepWell24 compared to a usual care control group. The investigators will conduct a pilot randomized controlled trial with participants randomly assigned to (1) SleepWell24; or (2) usual care for 60 days post-PAP prescription. The investigators will track recruitment/retention rates, app usage statistics, and measures of treatment satisfaction. The investigators will objectively measure PAP adherence to test whether the SleepWell24 group will have more hours/night of PAP usage compared to the usual care group. In an exploratory fashion, the investigators will also examine the effect of SleepWell24 on selected treatment outcomes (weight, daytime sleepiness, cognitive impairment, and health-related quality of life) and evaluate social cognitive and lifestyle behavior mediators of SleepWell24 on PAP adherence.

DETAILED DESCRIPTION:
This exploratory study will test the feasibility and initial efficacy of a mobile health smartphone intervention to increase adherence to positive airway pressure (PAP) therapy in newly diagnosed obstructive sleep apnea (OSA) patients treated at the Mayo Clinic Arizona Center for Sleep Medicine and associated outpatient clinics. This app, called SleepWell24, will include PAP adherence behavior change strategies (drawn from the evidence-based Sleep Apnea Self-Management Program), cloud-based linkages to a consumer-based PAP machine and wearable sensor that provides nightly feedback on PAP adherence and sleep and activity metrics, and a component to enhance patient-provider communication. The investigators will embed SleepWell24 within usual patient care at the Mayo Clinic Arizona Center for Sleep Medicine and associated outpatient clinics for app design/development, patient recruitment, and treatment feasibility/satisfaction. This design will ensure the best opportunity for clinical adoption. The primary aims are:

Aim 1: Determine the feasibility and acceptability of SleepWell24 from patient and provider perspectives.

Aim 2: Determine the extent to which SleepWell24 improves PAP adherence over the first 60 days of use relative to usual care.

As an exploratory aim the investigators will explore the effect of SleepWell24 on treatment outcomes (weight, daytime sleepiness, cognitive performance, health-related quality of life) and putative social cognitive and behavioral mediators of PAP adherence (e.g., self-efficacy, sleep quality, sedentary behavior, physical activity).

The investigators will test the feasibility, acceptability, initial efficacy and outcomes of SleepWell24 compared to usual care during the first 60 days of PAP use among 94 patients newly diagnosed with obstructive sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe obstructive sleep apnea diagnosed through clinical diagnostic testing and laboratory or home-based sleep study
* current use of appropriate Apple (iOS7 or higher) or Android (2.3 or higher) smartphone device
* Be able to read, write, and understand English
* Prescribed positive airway pressure therapy for obstructive sleep apnea

Exclusion Criteria:

* Do not agree to be randomized
* Currently participating in other lifestyle change programs
* Personal, health, cognitive, or psychological conditions that prevent full participation
* Pregnant, lactating, or trying to become pregnant
* Prescribed high-dose benzodiazepines
* Daily opioid medication use at night
* Unwilling to discontinue use of any current wearable sensor for the duration of the trial
* Unwilling to consent for out-of-pocket costs
* Previous treatment/referral for claustrophobia
* Previous Positive airway pressure therapy use
* Planning to travel for more than seven consecutive nights during the trial
* Currently engaging in shiftwork

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Recruitment and Retention | Duration of the trial (~60 days)
  numbers recruited and retained over the course of the trial
SleepWell24 application usage | Duration of the trial (~60 days)
  objective metrics of smartphone application usage by intervention group
Treatment acceptability/satisfaction | Baseline vs. Day 60 of trial
  Intervention acceptability questionnaire for both groups
Positive airway pressure therapy use | Duration of the trial (~60 days)
  How many hours per night therapy was used throughout the trial

SECONDARY OUTCOMES:
Body Mass Index | Baseline and follow-up visit between days 31 and 60
  body mass index according to weight and height
Daytime Sleepiness | Baseline, Day 30, Day 60 of trial
  Epworth Sleepiness Scale
Cognitive functioning | Baseline and follow-up visit between days 31 and 60
  Neurocognitive battery
Global Quality of Life due to physical and mental health via the Patient Reported Outcomes Measurement Information System Global Health Scale | Baseline, Day 30, Day 60 of trial
  The investigators will measure quality of life in general as informed by current physical and mental health using the quality of life in general as informed by current physical and mental health using the Patient Reported Outcomes Measurement Information System Global Health Scale. This Scale measures an individual's physical, mental, and social health, in general. This measure produces 2 scores: Physical Health and Mental Health. Summed raw scores are converted to T-score values with a mean of 50 and a standard deviation of 10. A higher T score indicates better Global Physical or Mental Health depending on the subscale used.
Sleep Apnea-Specific Quality of Life | Baseline, Day 30, Day 60 of trial
  The investigators will measure functional outcomes of sleep apnea with the Functional Outcomes of Sleep Questionnaire, which measures how difficult it is to carry out certain activities because of daytime sleepiness due to sleep apnea. It is a 10-item questionnaire representing 5 subscales. To obtain the total score, a mean-weighted item score is first computed for subscales with more than one item. Then the total score is derived by calculating the mean of the subscale scores and multiplying that mean by 5. Higher total scores indicate less difficulty with sleepiness due to sleep apnea affecting daytime activities. Scale ranges from 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Petrov, PhD, Principal Investigator — Arizona State University; Matthew Buman, PhD, Principal Investigator — Arizona State University
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Petrov ME, Epstein DR, Krahn L, Todd M, Park JG, St Louis EK, Morgenthaler TI, Hoffmann CM, Hasanaj K, Hollingshead K, Yu TY, Buman MP. SleepWell24, a Smartphone Application to Promote Adherence to Positive Airway Pressure Therapy: Feasibility and Acceptability in a Randomized Controlled Trial. Behav Sleep Med. 2024 Jul-Aug;22(4):420-432. doi: 10.1080/15402002.2023.2289442. Epub 2023 Nov 30. PMID 38032115